CLINICAL TRIAL: NCT06281756
Title: Cognitive Behavioral Therapy and Trazodone Effects on Sleep and Blood Pressure in Insomnia Phenotypes Based on Objective Sleep Duration: A Sequential Cohort/Randomized Controlled Trial
Brief Title: Cognitive Behavioral Therapy and Trazodone Effects on Sleep and Blood Pressure in Insomnia
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Alexandros Vgontzas, Professor, Department of Psychiatry, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00022285; 1UG3HL161342-01A1 (NIH)
Record Dates: First submitted 2024-02-19; First posted 2024-02-28 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Insomnia; Insomnia Chronic; Insomnia, Primary; Blood Pressure; Blood Pressure, High
Keywords: sleep; sleep disorder; insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Hypertension; Sleep Wake Disorders | interventions — Trazodone

STUDY DESIGN:
Intervention Model Description: A 4-site (Hershey, Pennsylvania; Pittsburgh, Pennsylvania; Denver, Colorado; and Quebec, Canada) cohort study will examine the effect of CBT-I as a recommended first-line treatment for insomnia. This will be followed by a placebo-controlled randomized controlled trial (RCT) in those who do not remit in the Cohort Study. The subsequent RCT will compare the efficacy of trazodone vs. placebo among CBT-I non-remitters.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Both prescribing physicians and participants will be blind to phenotype and treatment groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Subjects treated with Cognitive Behavior Treatment for Insomnia (CBT-I) with placebo (Placebo Comparator): Subjects with insomnia treated with Cognitive Behavior Treatment for Insomnia (CBT-I) for 8 weeks, then non-remitting subjects received placebo for 8 weeks.
  Interventions: Behavioral: Cognitive Behavioral Treatment for Insomnia (CBT-I); Other: Placebo
- Subjects treated with Cognitive Behavior Treatment for Insomnia (CBT-I) with Trazodone (Active Comparator): Subjects with insomnia treated with Cognitive Behavior Treatment for Insomnia (CBT-I) for 8 weeks, then non-remitting subjects received trazodone for 8 weeks.
  Interventions: Behavioral: Cognitive Behavioral Treatment for Insomnia (CBT-I); Drug: Trazodone

INTERVENTIONS:
Behavioral: Cognitive Behavioral Treatment for Insomnia (CBT-I) — Subjects will receive therapy for 8 weeks
Drug: Trazodone — Non-remitting subjects will receive Trazodone (dosage) for 8 weeks
  Arms: Subjects treated with Cognitive Behavior Treatment for Insomnia (CBT-I) with Trazodone
Other: Placebo — Non-remitting subjects will receive placebo for 8 weeks
  Arms: Subjects treated with Cognitive Behavior Treatment for Insomnia (CBT-I) with placebo

SUMMARY:
Individuals who have insomnia with short sleep duration (ISS) differ from individuals who have insomnia with normal sleep duration (INS) in terms of health risks (i.e., hypertension) and treatment response. This study will examine whether patients with ISS and INS demonstrate a differential response to two common insomnia treatments. One is behavioral, Cognitive Behavioral Therapy for Insomnia (CBT-I). The other is a widely prescribed, non-habit-forming medication, trazodone used at a low dose. The investigators' findings could lead to evidence-based treatment guidelines that help clinicians more effectively match treatments to insomnia patients and reduce associated health problems.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Able to read and effectively communicate in English at the United States sites or able to read and effectively communicate in English or French at the Canadian site.
* Meets criteria for chronic insomnia
* Body Mass Index (BMI) 18.5 kg/m2 and higher

Exclusion Criteria:

* Age < 18
* Unable to read and effectively communicate in English at the United States sites or able to read and effectively communicate in English or French at the Canadian site.
* Unwilling to share email address/cell phone number to accept survey links.
* Life time diagnosis of psychotic or bipolar disorder
* History of severe apnea or an Apnea Hypopnea Index (AHI) ≥15 that is not currently treated with Positive Airway Pressure (PAP) therapy, an oral device or an implanted device, or was not treated with surgery or weight loss.
* Started new or changed treatment for sleep apnea in the past three months
* Does not meet criteria for chronic insomnia
* Meets criteria for narcolepsy or hypersomnia disorder
* Meets criteria for circadian rhythm disorder (including night shift work)
* Unstable medical conditions that would make participation unsafe or unfeasible
* Falls resulting in hospitalization, significant injury or fracture within past 12 months
* 2 hospitalizations or emergency room visits within past 12 months for chronic conditions
* Active chemotherapy or radiation therapy for cancer
* Lifetime diagnoses/treatment of chronic renal failure, hepatic insufficiency, chronic heart failure
* Does not agree to refrain from other treatments for insomnia beyond what is offered in this study
* BMI less than 18.5
* Substance abuse or dependence in the past 12 months
* Current use of prescription or over the counter medications taken for sleep greater than 2 times per week
* Current use of systemic corticosteroids or opiate medications
* Current pregnancy or breastfeeding; plans to get pregnant or unwillingness to use birth control for the length of the study
* Current use of medications contraindicated with trazodone
* Sleep apnea or periodic leg movement disorder as determined by sleep study
* Blood Pressure levels defined as seated SBP greater than 180 or DBP greater than 110 mmHg
* EKG corrected QT interval greater than or equal to 500 ms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Remission of insomnia symptoms following Cognitive Behavioral Therapy for Insomnia (CBT-I) | 9 weeks
  Based on Insomnia Severity Index (ISI) published criteria; 0-28, with 0 being mild and 28 being severe
Remission of insomnia symptoms following trazodone/placebo Randomized Controlled Trial (RCT) | 9 weeks
  Based on Insomnia Severity Index (ISI) published criteria; 0-28, with 0 being mild and 28 being severe
Remission of insomnia symptoms 6 months following completion of CBT-I Or RCT Treatment | 35 weeks
  Based on Insomnia Severity Index (ISI) published criteria; 0-28, with 0 being mild and 28 being severe

SECONDARY OUTCOMES:
Insomnia Severity Index (ISI) Score following CBT-I | 9 weeks
  0-28, with 0 being mild and 28 being severe
Polysomnography (PSG) Sleep efficiency following Cognitive Behavioral Therapy for Insomnia (CBT-I) | 9 weeks
  Polysomnography (PSG) Sleep efficiency measured as a percentage of time asleep during sleep study
Actigraphy Sleep efficiency following Cognitive Behavioral Therapy for Insomnia (CBT-I) | 9 weeks
  Actigraphy Sleep efficiency measured as estimated sleep time at home (2 week period)
Evening Cortisol levels following CBT-I | 9 weeks
  Cortisol levels measured in saliva collected following CBT-I
Insomnia Severity Index (ISI) Score following RCT | 9 weeks
  0-28, with 0 being mild and 28 being severe
PSG Total Sleep Time (TST) following RCT | 9 weeks
  PSG Total Sleep Time measured in minutes asleep during sleep study following RCT
Actigraphy Total Sleep Time (TST) following RCT | 9 weeks
  Actigraphy Total Sleep Time measured in minutes asleep during home study following RCT
Home Blood Pressure (HBP) Morning Systolic Blood Pressure (SBP) | 9 weeks
  Morning SBP Blood Pressure Readings measured at home (7 day period)
Home Blood Pressure (HBP) Morning Diastolic Blood Pressure (DBP) | 9 weeks
  Morning DBP Blood Pressure Readings measured at home (7 day period)
Evening Cortisol levels following RCT | 9 weeks
  Cortisol levels measured in saliva collected following RCT
Evening Cortisol levels 6 months following completion of CBT-I or RCT Treatment | 35 weeks
  Cortisol levels measured in saliva 6 months following CBT-I Or RCT Treatment

CONTACTS AND LOCATIONS:
Overall Officials: Alexandros Vgontzas, MD, Principal Investigator — Professor, Psychiatry
Locations (4):
- United States (3):
  - National Jewish Health, Denver, Colorado
  - Penn State University, Hershey, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
- Université Laval, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
The investigators have extensive experience preparing data and documentation to be available for public. They agree to abide by the principles for sharing research resources described by the National Heart, Lung, Blood Institute (NHLBI). A copy of the data will be uploaded to the NHLBI Biologic Specimen and Data Repositories Information Coordinating Center (BioLINCC) repository. The datasets will not include any personal identifiers related to participants or clinical sites. Dates will be de-identified through a date-shifting algorithm to mask actual dates while maintaining a relation to the epoch in which events occurred. Data tables will be exported in comma-separated format, readable by statistical software. Variable dictionaries and code books, detailing variable description, format, value domain and labels, will be produced. Raw data files for polysomnogram/actigraphy/cortisol will also be made available, ensuring that data are linkable to study data and data are de-identified.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Data collected for aim 1 (an observational study) and aim 2 (a randomized clinical trial) will be made available no more than 3 years after the completion of the last follow-up assessment. Data will be submitted to the Program Officer and uploaded to the NHLBI BioLINCC repository no later than 3 years after the end of clinical activity or 2 years after the main outcomes paper is published, whichever comes first.
Access Criteria: NHLBI BioLINCC repository
URL: https://biolincc.nhlbi.nih.gov/home/